CLINICAL TRIAL: NCT01239628
Title: A National, Prospective, Non-interventional Survey to Evaluate Injection Intervals and Treatment Modalities up to 3 Years Follow up of Botulinum Toxin A in Adult Subjects Suffering From Upper Limb Spasticity Post-CVA (Cerebrovascular Accident)
Brief Title: A Prospective, Non-interventional Survey to Evaluate Injection Intervals and Treatment Modalities of Botulinum Toxin A (BoNT-A) in Adult Patients Suffering From Upper Limb Spasticity After Stroke
Acronym: DECIDE
Status: Terminated | Type: Observational
Why Stopped: Participant enrolment was lower than expected
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-48-52120-152
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Upper Limb Spasticity After Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the protocol is to evaluate injection intervals and treatment modalities up to 3 years follow-up of botulinum toxin A (BoNT-A) in adult patients suffering from upper limb spasticity after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Subject able to comply with the protocol
* Provision of written informed consent prior to collecting the data
* Male or female patients of 18 years or older
* Presenting with upper limb spasticity after stroke for which treatment with botulinum toxin A is indicated

Exclusion Criteria:

* The subject has already been included in this survey
* Patients who already received BoNT-A treatment for upper limb spasticity
* Patients with known intolerance for BoNT-A
* Subjects unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a history of stroke, suffering from upper limb spasticity
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2010-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Documentation of the injection intervals | 3 years
Documentation of treatment modalities | 3 years

SECONDARY OUTCOMES:
Documentation of the main reason(s) for change in injection intervals | 3 years
Documentation of the main reason(s) for dose change(s) | 3 years
Documentation of the patient satisfaction with the treatment | 3 years
Documentation of the physician satisfaction with the treatment | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Neurology, Study Director — Ipsen
Locations (11):
- Belgium (11):
  - St- Augustinus, Antwerp
  - ZNA Middelheim, Antwerp
  - AZ St-Jan, Bruges
  - RevalidatieZiekenhuis RevArte, Edegem
  - AZ Sint Lucas, Ghent
  - Revalidatiecentrum St Ursula, Herk-de-Stad
  - ZOL, Campus Sint Barbara, Lanaken
  - Heilig Hart Ziekenhuis, Lier
  - Hôpital Marie Curie, Lodelinsart
  - CHU Leonardo da Vinci, Montigny-le-Tilleul
  - CHPLT Peltzer, Verviers